CLINICAL TRIAL: NCT02835703
Title: Clinical Assessment of Perfusion Techniques During Surgical Repair of Coarctation of Aorta With Aortic Arch Hypoplasia in Infants
Brief Title: Clinical Assessment of Perfusion Techniques During Repair of Coarctation With Aortic Arch Hypoplasia in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTAAR
Record Dates: First submitted 2016-07-06; First posted 2016-07-18 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Coarctation of Aorta
Keywords: Congenital heart disease; Coarctation of aorta; Aortic arch hypoplasia; Cerebral selective antegrade perfusion; Double arterial cannulation
MeSH Terms: conditions — Aortic Coarctation; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Deep hypothermic arrest (Active Comparator): Surgical repair of coarctation of aorta under deep hypothermic circulatory arrest
  Interventions: Procedure: Surgical repair of coarctation of aorta
- Selective antegrade cerebral perfusion (Active Comparator): Surgical repair of coarctation of aorta using selective antegrade cerebral perfusion
  Interventions: Procedure: Surgical repair of coarctation of aorta
- Double arterial cannulation (Active Comparator): Surgical repair of coarctation of aorta using cerebral antegrade perfusion with descending aortic cannulation
  Interventions: Procedure: Surgical repair of coarctation of aorta

INTERVENTIONS:
Procedure: Surgical repair of coarctation of aorta — Surgical repair of coarctation of aorta with aortic arch hypoplasia under CPB

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of three main perfusion methods in surgical repair of coarctation of aorta with aortic arch hypoplasia in infants.

DETAILED DESCRIPTION:
Three perfusion techniques of visceral protection will be assessed - deep hypothermic circulatory arrest, selective antegrade cerebral perfusion and double arterial cannulation (perfusion of brachiocephalic artery with thoracic descending aorta by two arterial cannulas)

ELIGIBILITY:
Inclusion Criteria:

* coarctation with severe aortic arch hypoplasia (distal aortic arch z-score < -2)
* coarctation of aorta with septal defects

Exclusion Criteria:

* coarctation with mild aortic arch hypoplasia (distal aortic arch z-score > -2)
* complex congenital heart diseases including aortic arch hypoplasia (e.g. transposition of great arteries, double oulet right ventricle, atrioventricular septal defect, Shone's complex)
* univentricular and duct-dependent heart defects
* aortic valve and/or mitral valve stenosis/hypoplasia (aortic valve or mitral valve z-score < -2.0)
* left ventricular dysfunction (left ventricle ejection fraction < 60%)
* congenital renal or central nervous system anomalies
* related infectious diseases
* prematurity (gestational age < 37 weeks)

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events in early postoperative period | 30 days after surgery
  Number of participants with adverse events that are related to treatment (including hospital mortality, renal injury (pRIFLE criteria), neurological complications (confirmed by CT or MRI) )

SECONDARY OUTCOMES:
Degree of inotropic support (inotropic score) | through ICU stay, an average of 3 weeks
Intraoperative blood loss (ml) | intraoperatively
Temperature of cooling (C) | intraoperatively
Duration of CPB (min) | intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kulyabin YY, Bogachev-Prokophiev AV, Soynov IA, Omelchenko AY, Zubritskiy AV, Gorbatykh YN. Clinical Assessment of Perfusion Techniques During Surgical Repair of Coarctation of Aorta With Aortic Arch Hypoplasia in Neonates: A Pilot Prospective Randomized Study. Semin Thorac Cardiovasc Surg. 2020 Winter;32(4):860-871. doi: 10.1053/j.semtcvs.2020.04.015. Epub 2020 May 22. PMID 32446921